CLINICAL TRIAL: NCT00787423
Title: Developing Field Tools for Real-Time Assessment of Exposure to Psychosocial Stress and Drug Use in an Outpatient Treatment Population
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909020; 09-DA-N020
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-05-06

CONDITIONS: Stress; Drug Abuse
Keywords: Field Tools; Stress; Ecological Monetary Assessment (EMA); Global Positioning Units; Natural History; Psychosocial Stress
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COHORT 1: Individuals from 18 to 75 years of age who are current heroin users seeking treatment for addiction and who spend most of their time in Baltimore city.

SUMMARY:
Background:

- Researchers are interested in developing more accurate methods to assess environmental influences on psychological stress and drug use. One key to a more accurate assessment of environmental influences is minimizing the delay between exposure and reporting. Portable devices such as personal digital assistants (PDAs) and global positioning system (GPS) units may be able to provide a more real-time image of these factors.

Objectives:

- To assess the use of PDAs to measure stress and drug use, and GPS units to assess the effects of neighborhood environment in an outpatient treatment population.

Eligibility:

* Individuals from 18 to 75 years of age who are current heroin users seeking treatment for addiction and who spend most of their time in Baltimore city.
* Participants must be able to visit the research and treatment center at least three times per week for regular tests.

Design:

* Participants will be in the study for approximately 28 weeks (7 months).
* A series of three laboratory session examining responsiveness to standardized stressors will occur both early in treatment and will be repeated late in treatment.
* Participants will undergo 18 weeks of daily methadone maintenance. Urine samples will be collected three times weekly.
* To track drug use, stress, and geographical location (a measure of environmental risk), each participant will carry a PDA and a GPS unit for 16 of the 18 weeks. Participants will make entries (1) each time that they use a drug and (2) each time they feel overwhelmed, anxious, or stressed more than usual. Participants will also make three random-signal-triggered recordings per day and one brief (end of day) recording.
* Retrospective self-report questionnaires on drug use and stress will be given regularly.
* After 18 weeks of methadone maintenance, participants will discontinue carrying the PDA and GPS unit and will have the choice of transferring to a community clinic or undergoing a 10-week taper from methadone at the research clinic. Participants who stay for the taper will continue to provide urine samples, but only once a week.

DETAILED DESCRIPTION:
Background. This protocol arose in response to NIH s Genes and Environment Initiative (GEI). There is no genetic component to this protocol (update: no genetics initially but added by amendment in February 2013); rather, the goal is to develop field-deployable measures of environmental influences (stressors, drug exposure, etc.) that can ultimately be used in studies of gene-environment interactions.

<TAB>

Objective. To use smartphones as electronic diaries (EDs) and passive data collection tools to measure geographical location, physical activity, social interactions, stress and drug use; Global Positioning System (GPS) units to assess geographical location; biological samples for genetic testing; Daysimeters and Dimesimeters to assess circadian rhythm; AutoSense and Health Tag to collect ambulatory physiological and activity data in real time; social media language to assess content associated with stress and drug use; and to assess the feasibility and acceptability of mobile HIV/STD Risk Reduction (HIVRR) or stress-reduction intervention with feedback from Health Tag delivered via ED in real time.

Participant population. Opioid-dependent outpatient adults (up to 500 enrolled; up to 400 completers). Target enrollment will include 40% women and 60% minorities (mostly African-American).

Experimental design. A natural-history study of stress (both personal and environmental) and drug use.

Methods. Participants will undergo 22 weeks of Office-based Opiate Treatment (OBOT) at Archway clinic or methadone or buprenorphine/naloxone (henceforth buprenorphine ) maintenance elsewhere, and will be offered at least 8 weeks of methadone or buprenorphine taper (weeks 23-30). OBOT buprenorphine will be administered twice weekly in the clinic, with additional doses given to take at home. Social media language will be collected at baseline and weekly during the study. To track drug use, stress, physical activity, social interactions, and geographical location (a measure of environmental risk), each participant will carry an ED and a GPS unit or wireless smartphone for up to 16 weeks. Event-triggered entries will be initiated by participants (1) each time that they use a drug and (2) each time they feel overwhelmed, anxious, or stressed more than usual. Participants will also make 3 random-signal-triggered recordings per day and one brief end of day recording. We will compare these ecological momentary assessment (EMA) results with more traditional assessments of drug use and stress: (1) urine will be collected two or three times weekly during weeks 1-22 and once weekly during the optional methadone or buprenorphine taper (weeks 23-30), (2) retrospective self-report questionnaires on drug use and stress will be given regularly, and (3) laboratory session examining responsiveness to a standardized stressor will occur during the 4th -6th week. Blood draws and anthropometric measurements to assess allostatic load (a physiological marker of long-term cumulative stress) and blood samples will be obtained for genetic analysis during the 2nd -4th week. After week 12, we will also assess the impact of opioid agonist treatment on the hypothalamic-pituitary-adrenal (HPA) axis which is involved in modulating stress. After 18 weeks of opioid agonist maintenance, participants will begin an additional 4 weeks of maintenance, during which they will not carry the wireless smartphone or ED and GPS unit unless they are participating in a secondary study that includes those measures. At the end of 22 weeks, participants will have the choice of transferring to a community clinic or undergoing an eight-week taper at the Archway clinic. Individuals receiving treatment in other programs may participate in the treatment elsewhere arm of the study. In this arm, ED and GPS data will be collected for 8 weeks; urine drug screens will be collected three times weekly. Secondary studies: Up to 70 participants will be asked to wear the Daysimeter and an Actigraph activitymonitor wristwatch for 18 days (two 72-hour intervals repeated three times) and the Dimesimeter daily (24 hours/day) for 16 weeks (completed September 2015). Up to 80 participants will be asked to wear the AutoSense for four 1-week periods, including during laboratory sessions. Up to 40 participants will be enrolled in the mHIVRR evaluation program for 4 weeks during the Maintenance Phase (completed October 2013). Up to 100 participants will be asked to wear a SleepProfiler during 7 nights to assess sleep architecture (completed March 2019). Up to 50 participants will be asked to wear the Health Tag for up to 6 weeks.

Primary outcome measures: (1) EMA reports of drug use and psychosocial stress, and (2) real-time assessment of environmental risk exposure as measured via integration of GPS data with neighborhood psychosocial indicators. Data for the methadone and buprenorphine groups will be analyzed separately for the primary outcome measures and combined as appropriate.

Secondary outcome measures: To determine the feasibility and acceptability of using (1) the Daysimeter/Dimesimeter and Actigraph to collect real-time field data on light exposure and its impact on circadian rhythms, and (2) the Autosense to collect real-time field data on physiological function. Also, to (3) combine Daysimeter/Dimesimeter data with electronic-diary data to determine whether heroin/cocaine users experience circadian disruption and, if so, how this disruption is related to psychosocial stress and illicit drug use, (4) combine Autosense data with electronic-diary data to determine if physiological responses to triggers can be used to inform drug relapse prevention efforts, (5) To determine the feasibility and acceptability of interactive mHIVRR software programs to deliver counseling and HIV education, and to determine whether they reduce HIV-related risk via increased HIV/STD knowledge, (6) to determine if the HPA axis is normal after at least 3 months of opioid agonist treatment, (7) to incorporate genetic characteristics as predictors of EMA and GMA data and other behavioral measures, (8) to assess how objectively measured sleep quality is associated with EMA-reported psychosocial stress and reward responsiveness, and with geographical exposure to stressful and rewarding environments, (9) to determine the feasibility of using a more up-to-date EMA interface and device, and to examine the relationship between opioid withdrawal symptoms and successful taper from methadone or buprenorphine maintenance and (10) to obtain qualitative data on participants perceptions of their environments, in order to inform future work and to help explain why participants seem to do better in more disordered environments. (11) To evaluate the feasibility of using the Spire Health Tag to infer emotional state from respiratory status, with the eventual goal (not an aim in this protocol) of providing a just-in-time intervention to relieve stress and anxiety. (12) to determine the feasiblilty of using passively collected smartphone data to assess physical activity and social interactions to infer daily behaviors, such as physical movement (activity, mobility patterns) and social interactions (computer-mediated communications), (13) to describe and analyze differences in the frequency and content of dialogue on social media to determine the words or phrases associated with drug use; drug treatment; recovery; and risk and protective factors for drug use (e.g., stress levels, anxiety, depression, social support).

ELIGIBILITY:
* INCLUSION CRITERIA:

Daily Treatment and OBOT arm-

Participants will be eligible for inclusion in the study if they meet the following criteria:

1. Age between 18 and 75
2. Physical dependence on opioids (by positive urine and/or frank opioid withdrawal)
3. Baltimore City or Baltimore, Harford, Howard, or Anne Arundel County home address or report of working in Baltimore city or spending most of their waking hours in Baltimore city.

Treatment Elsewhere (TE) arm-

Participants will be eligible for inclusion in the study if they meet the following criteria:

1. age between 18 and 75;
2. Receiving methadone or buprenorphine treatment for opioid dependence at a community substance abuse treatment program;
3. Baltimore City or Baltimore, Harford, Howard, or Anne Arundel County home address or report of working in Baltimore city or spending most of their waking hours in Baltimore city.

EXCLUSION CRITERIA:

Daily Treatment and OBOT arm-

1. History of any DSM-IV psychotic disorder; history of bipolar disorder; current Major Depressive Disorder;
2. current dependence on alcohol or sedative-hypnotic, e.g. benzodiazepine (by DSM-IV criteria);
3. cognitive impairment severe enough to preclude informed consent or valid self-report;
4. Any condition that interferes with urine collection;
5. medical illness (e.g., cirrhosis, nephrotic syndrome, thyroid disease, ischemic heart disease, epilepsy, panhypopituatarism, adrenal insufficiency, etc.) or medications that, in the view of the investigators, would compromise participation in research (e.g., glucocorticoids, adrenal extract supplements, spirnolactone, pregnenolone, etc.)

Treatment Elsewhere (TE) arm-

1. History of any DSM-IV psychotic disorder; history of bipolar disorder; current Major Depressive Disorder;
2. cognitive impairment severe enough to preclude informed consent or valid self-report;
3. Any condition that interferes with urine collection.

Further exclusions and rescheduling criteria for all laboratory sessions-

* The self-reported use of over-the-counter or as needed medications (e.g., antacids, sleeping aids, antihistamines, etc.) for 5 days prior to the scheduled session
* Positive breathalyzer test (BAL > 0) and/or acute intoxication from illicit drugs or alcohol
* Positive pregnancy test
* Self-report of recent pregnancy or child birth (and no resumption of normal menses)
* Failure to fast.

Participants will be allowed to reschedule 1 time (in total, for the 2 sessions).

* Other reasons for which participants may be rescheduled:
* They report significant recent health (e.g. influenza, infection, wound) or emotional (e.g. death in the family) events.
* Are late for session

Further inclusion/exclusion for the HPA axis component-

Inclusion

* Receiving buprenorphine agonist therapy (dose range 16-24 mg)
* Stable buprenorphine dose for 30 days prior

Exclusions (based on impact on HPA axis and neuroendocrine function)

* HIV+
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Opioid-dependent outpatient adults (up to 500 enrolled; up to 400 completers). Target enrollment will include 40% women and 60% minorities (mostly African-American).@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 373 (Actual)
Dates: Start 2009-07-14 (Actual)

PRIMARY OUTCOMES:
Real-time assessment of environmental risk exposure as measured via integration of GPS data with the Neighborhood Psychosocial Index | real-time assessment
  Real-time assessment of environmental risk exposure as measured via integration of GPS data with the Neighborhood Psychosocial Index
EMA reports of drug use and psychosocial stress | real-time assessment
  EMA reports of drug use and psychosocial stress

SECONDARY OUTCOMES:
To determine the feasibility and acceptability of interactive mHIVRR software programs to deliver counseling and HIV education, and to determine whether they reduce HIV-related risk via increased HIV/STD knowledge | Ongoing
  To determine the feasibility and acceptability of interactive mHIVRR software programs to deliver counseling and HIV education, and to determine whether they reduce HIV-related risk via increased HIV/STD knowledge
To evaluate sleep quality in relationship to drug use and stress exposure | Ongoing
  To evaluate sleep quality in relationship to drug use and stress exposure
Incorporate genetic characteristics as predictors of EMA and GMA data and other behavioral measures | Ongoing
  Incorporate genetic characteristics as predictors of EMA and GMA data and other behavioral measures
To determine if the HPA axis is normal after at least 3 months of opioid agonist treatment | Ongoing
  To determine if the HPA axis is normal after at least 3 months of opioid agonist treatment
Determine the feasibility of using a more up-to-date EMA interface and device | Ongoing
  Determine the feasibility of using a more up-to-date EMA interface and device
To assess how objectively measured sleep quality is associated with EMA-reported psychosocial stress and reward responsiveness, and with geographical exposure to stressful and rewarding environments | Ongoing
  To assess how objectively measured sleep quality is associated with EMA-reported psychosocial stress and reward responsiveness, and with geographical exposure to stressful and rewarding environments
Accuracy and helpfulness of the Health Tag | Ongoing
  Accuracy and helpfulness of the Health Tag
Combine Autosense data with electronic-diary data to determine if physiological responses to triggers can be used to inform drug relapse prevention efforts | Ongoing
  Combine Autosense data with electronic-diary data to determine if physiological responses to triggers can be used to inform drug relapse prevention efforts
Combine Daysimeter/Dimesimeter data with electronic-diary data to determine whether heroin/cocaine users experience circadian disruption and, if so, how this disruption is related to psychosocial stress and illicit drug use | Ongoing
  Combine Daysimeter/Dimesimeter data with electronic-diary data to determine whether heroin/cocaine users experience circadian disruption and, if so, how this disruption is related to psychosocial stress and illicit drug use
Feasibility and acceptability of using the Autosense to collect real-time field data on physiological function | Ongoing
  Feasibility and acceptability of using the Autosense to collect real-time field data on physiological function
Feasibility and acceptability of using the Daysimeter/Dimesimeter and Actigraph to collect real-time field data on light exposure and its impact on circadian rhythms | Ongoing
  Feasibility and acceptability of using the Daysimeter/Dimesimeter and Actigraph to collect real-time field data on light exposure and its impact on circadian rhythms
To determine the feasibility of using passively collected smartphone data to assess physical activity and social interactions to infer daily behaviors, such as physical movement (activity, mobility patterns) and social interactions (computer-med... | Ongoing
  To determine the feasibility of using passively collected smartphone data to assess physical activity and social interactions to infer daily behaviors, such as physical movement (activity, mobility patterns) and social interactions (computer-mediated communications)
To describe and analyze differences in the frequency and content of dialogue on social media to determine the words or phrases associated with drug use; drug treatment; recovery; and risk and protective factors for drug use (e.g., stress levels,... | Ongoing
  To describe and analyze differences in the frequency and content of dialogue on social media to determine the words or phrases associated with drug use; drug treatment; recovery; and risk and protective factors for drug use (e.g., stress levels, anxiety, depression, social support).

CONTACTS AND LOCATIONS:
Overall Officials: Brenda L Curtis, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
The protocol does not address IPD activities.

REFERENCES:
- [Background] Boardman JD, Finch BK, Ellison CG, Williams DR, Jackson JS. Neighborhood disadvantage, stress, and drug use among adults. J Health Soc Behav. 2001 Jun;42(2):151-65. PMID 11467250